CLINICAL TRIAL: NCT07038200
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous AOC 1020 for the Treatment of Facioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: A Study to Evaluate Del-brax (Also Referred to as AOC 1020) in Participants With FSHD
Acronym: FORTITUDE-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOC 1020-CS3
Record Dates: First submitted 2025-06-13; First posted 2025-06-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Facioscapulohumeral Muscular Dystrophy; FSHD; FSHD - Facioscapulohumeral Muscular Dystrophy; FSHD1; FSHD2; Fascioscapulohumeral Muscular Dystrophy; Fascioscapulohumeral Muscular Dystrophy Type 1; Fascioscapulohumeral Muscular Dystrophy Type 2; Facioscapulohumeral Muscular Dystrophy 1; Facioscapulohumeral Dystrophy; Facio-Scapulo-Humeral Dystrophy; Facioscapulohumeral Muscular Dystrophy 2; Facioscapulohumeral Muscular Dystrophy Type 1 (FSHD1); FSH Muscular Dystrophy; Landouzy Dejerine Dystrophy; Landouzy-Dejerine Muscular Dystrophy; Landouzy-Dejerine Syndrome
Keywords: Avidity; Avidity Biosciences; del-brax; del brax; delbrax; AOC1020; AOC 1020; delpacibart braxlosiran; FORTITUDE-3; FORTITUDE Phase 3; FORTITUDE; FORTITUDE 3
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Facioscapulohumeral Muscular Dystrophy 1B; Facioscapulohumeral muscular dystrophy 1a | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- del-brax (Experimental): Del-brax (AOC 1020) will be administered 13 times
  Interventions: Drug: AOC-1020
- placebo (Placebo Comparator): Saline will be administered 13 times
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AOC-1020 — Placebo
  Other Names: del-brax
  Arms: del-brax
Drug: Placebo — Placebo will be administered by intravenous (IV) infusion.
  Other Names: saline
  Arms: placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous AOC 1020 for the Treatment of Facioscapulohumeral Muscular Dystrophy (FSHD)

DETAILED DESCRIPTION:
The study consists of a Screening Period of up to 6 weeks and 72-week Treatment Period. The anticipated duration is approximately 78 weeks.

Participants will be randomized to receive an intravenous infusion of either del-brax or placebo at the clinical study site every 6 weeks for a total of 13 doses. The final dose will occur at Week 72, followed by a final assessment at Week 78.

After completion of the Week 78 visit, eligible participants will have the option to enroll into an open label extension (OLE) study, pending regulatory approval. Participants who decline participation in the OLE will be followed for a period of 12 weeks for safety.

An Independent Data Monitoring Committee (IDMC) comprising members independent and external to the Sponsor will review safety, tolerability, and efficacy (as needed) data of this study at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and genetic diagnosis of FSHD1 or FSHD2
* Ability to walk independently at pre-specified walking speed (orthoses and ankle braces allowed) for at least 10 meters at screening
* Adequate muscle strength based on QMT composite score

Exclusion Criteria:

* Breastfeeding, pregnancy, or intent to become pregnant during the study
* Unwilling or unable to comply with contraceptive requirements
* Abnormal lab values, conditions or diseases that would make the participant unsuitable for the study
* Blood Pressure > 140/90 mmHg at Screening
* Treatment with another investigational drug or biological agent within 1 month of Screening or 5 half-lives of the drug, whichever is longer
* Treatment with an oligonucleotide within 9 months of Screening

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Quantitative Muscle Testing (QMT) composite score | Baseline through Week 78

SECONDARY OUTCOMES:
10-Meter Walk/Run Test (10MWRT) | Baseline through Week 78
Timed Up-and-Go (TUG) | Baseline through Week 78
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Item Bank v2.0-Physical Function-Short Form 20a Questionnaire | Baseline through Week 78
Worst Pain Numeric Rating Scale (NRS) | Baseline through Week 78
Patient Global Impression of Severity/Change (PGI-S/PGI-C) | Baseline through Week 78
DUX-4 Regulated Circulating Biomarker of FSHD Disease Biology | Baseline through Week 78
Circulating Creatine Kinase (CK) | Baseline through Week 78

CONTACTS AND LOCATIONS:
Locations (22):
- United States (14):
  - University of California Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (4):
  - University of Calgary - Cumming School of Medicine, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Genge Partners Inc, Montreal, Quebec
- Japan (4):
  - National Hospital Organization Osaka Toneyama Medical Center, Osaka
  - The University of Osaka Hospital, Osaka
  - National Hospital Organization Sendai Nishitaga Hospital, Sendai
  - National Center of Neurology and Psychiatry, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.aviditybiosciences.com/
- See also: Related Info — https://www.forwardstudy.com/